CLINICAL TRIAL: NCT02127762
Title: The Effect of an Inter-Disciplinary Program, Including Mindfulness Based Stress Reduction, on Psychosocial Function, Pain and Metabolism in Patients With Painful Diabetic Peripheral Neuropathy
Brief Title: The Effect of Mindfulness Based Stress Reduction in Patients With Painful Diabetic Peripheral Neuropathy
Acronym: AWARE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Canadian Diabetes Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 20120541-01H; # OG-2-12-3722-HN (Other Grant/Funding Number: Canadian Diabetes Association Grant)
Record Dates: First submitted 2014-04-29; First posted 2014-05-01 (Estimated); Last update posted 2018-06-13 (Actual); Status verified 2018-06

CONDITIONS: Diabetes Mellitus; Type I Diabetes; Type II Diabetes; Diabetic Peripheral Neuropathy; Chronic Pain
Keywords: Pain; Quality of Life; Glycemic Control; diabetic neuropathy; mindfulness; stress reduction; adult; chronic pain; depression; cortisol
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Chronic Pain; Pain; Diabetic Neuropathies; Depression | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mindfulness Based Stress Reduction (Experimental): Participants assigned to this group will be enrolled in an Mindfulness-Based Stress Reduction (MBSR) program following medical treatment optimization. The MBSR program will be composed of eight weekly 2.5 hour sessions and one 6 hour session midway through the course.
  Interventions: Behavioral: Mindfulness Based Stress Reduction
- Wait-listed Control Group (No Intervention): Participants assigned to this group after medical treatment optimization will act as wait-list controls for the MBSR group. They will be enrolled in the MBSR workshop 3 months after the corresponding intervention group completes the program.

INTERVENTIONS:
Behavioral: Mindfulness Based Stress Reduction — Consists of eight weekly 2.5 hour sessions and one 6 hour session midway through the course. All sessions will be conducted by a psychologist or social worker with experience in chronic pain, formal MBSR training and 5 years of experience leading MBSR groups.
  Arms: Mindfulness Based Stress Reduction

SUMMARY:
By 2020, it is estimated that 3.7 million Canadians will have diabetes mellitus, with type 2 diabetes (T2DM) accounting for more than 90% of cases. Estimates of the prevalence of diabetic peripheral neuropathy among adults with T2DM range from 26% to 47%. It increases with patient age and duration of disease and it can be as high as 60 to 70% in older cohorts. Diabetic peripheral neuropathy is documented in most studies as numbness, tingling, pain and/or objective sensory changes. Pain is an early manifestation of neuropathy and may be the presenting symptom of diabetes. Even the best medications and procedures rarely relieve more than 30% of the discomfort of chronic painful conditions. Diabetic patients continue to experience debilitating and disabling pain. Pain affects our ability to work, our ability to participate in recreational activities, our mood and our relationships. It is well-established that an interdisciplinary approach is key to the treatment of some types of chronic pain, but little research has been done on the effectiveness of interdisciplinary treatments for patients suffering from painful diabetic peripheral neuropathy. The investigators will evaluate the effectiveness of an interdisciplinary approach combining medical treatment and mindfulness-based stress reduction (MBSR) to reduce disability and improve quality of life among patients with painful diabetic peripheral neuropathy. The investigators will also evaluate the impact of the program on psychological distress, pain cognitions, and biomarkers of stress and glycemic function.

DETAILED DESCRIPTION:
The investigators will recruit 110 adults with painful diabetic peripheral neuropathy. All will have their medical treatment optimized by a pain medicine specialist before being randomly assigned to either an 8-week group MBSR program or a wait-list. All participants will complete self-report questionnaires, provide a hair sample for cortisol measurements and a blood sample to measure glycemic index. We will be collecting outcome data for both groups. Patients randomized to MBSR will have data collected at 4 time points: 1) before medical optimization; 2) after medical optimization and before the MBSR group intervention begins, 3) 2 weeks after the group intervention; and 4) 3 months following completion of MBSR. Patients randomized to control will have data collected at 6-7 time points depending on when are participants enrolled in the trial: 1) before medical optimization; 2) after medical optimization and before the MBSR group intervention begins; 3) 2 weeks after the group intervention; 4) 3 months following completion of MBSR; 5) Re-test before control group intervention begins; 6) 2 weeks after control group intervention; and 7) 3 months after control group intervention.

The primary hypothesis is that after all patients are medically optimized, those randomized to MBSR will have a 30% higher incidence of clinically significant (≥1.0 decrease in mean BPI interference score) improvement (responders) compared to controls measured 3 months following completion of MBSR. A significant change is defined as ≥ 1 decrease in BPI interference score. A one point change on the Interference Scale, has been recommended by the Initiative on Methods, Measurement, and Pain Assessment in Clinical Trials (IMMPACT) group as a minimally clinically important change. This design controls for the effect of time and disease fluctuation, regression to the mean, and the effect of testing. In this preliminary research, where our primary goal is to establish proof of concept and obtain data needed to plan a comparative trial, we are not controlling for the placebo effect. We believe that a wait-list controlled study is the necessary foundation on which to build a rigorous program of research.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged > 18 years
* Type 1 or Type 2 Diabetes Mellitus (receiving insulin or not)
* HbA1c 6.5%-9.9%
* Diagnosis of Diabetic Peripheral Neuropathy (DPN) > 1 year
* Report of pain > 6 months
* Score >3 on Douleur Neuropathique-4 Questionnaire
* VAS completed 5/7 days; Average VAS score >4 and <9 (i.e., moderate to severe pain).
* Ability to attend a minimum of 7 of 9 MBSR workshops

Exclusion Criteria:

* Peripheral vascular disease requiring revascularization of lower limb or amputation
* Pregnant or lactating
* Active alcohol or drug abuse/dependence
* Previous MBSR training
* Co-morbidity preventing assessment or understanding of questionnaires
* Inability to speak English or French

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2012-09; Primary Completion 2016-06 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Change from baseline in pain-related disability, as measured by the Brief Pain Inventory. Pain interference scale at 3-month post-intervention. | Baseline and 3 months post-intervention
  The primary outcome is pain-related disability, as measured by the Brief Pain Inventory pain interference scale which consists of 7 numerical scales (0 to10) rating pain interference with general activity, mood, walking ability, work, relations with other people, sleep and enjoyment of life.

SECONDARY OUTCOMES:
Change from baseline in pain severity, as measured by the Brief Pain Inventory - Pain Severity scale, at 3 months post-intervention | Baseline and 3 months post-intervention
  Pain Severity will be measured using the Brief Pain Inventory (BPI) - Pain Severity. The BPI consists of 4 numerical scales (0 to 10) rating pain severity at its worst, at its least, on average, and at the time of filling out the measure. Each severity question is analyzed individually.
Change from baseline in mood states, as measured by the Profile of Mood States scale, at 3 months post-intervention. | Baseline and 3 months post-intervention
  The Profile of Mood States (POMS-2A) will be used to measure mood disturbance. Participants are asked to rate 65 adjectives using a 5-point likert scale (0= not at all, to 4 = extremely) based on how they have been feeling during the past week, including the day they are filling out the questionnaire. A total mood disturbance score is calculated, as well as scores for 6 subscales: depression, tension-anxiety,anger-hostility, vigor-activity, fatigue, confusion-bewilderment.
Overall change in status from baseline, as measured by Patient Global Impression of Change scale, at 3 months post-intervention. | Baseline and 3 months post-intervention
  The participants perceived degree of change in overall status will be measured using the Patient Global Impression of Change (PGIC) scale. The PGIC uses a 7-point likert scale (very much worse, to very much better) to measure how much the participant feels their overall status has changed since the start of the study.
Change from baseline in stress, as measured by the Perceived Stress Scale, at 3 months post-intervention. | Baseline and 3 months post-intervention
  The Perceived Stress Scale (PSS) will be used to measure the participants' perceived stress levels. The PSS uses a 5-point likert scale (0=Never, to 4=Very often) to measure the degree of stress a participant has experienced over the past month. A total perceived stress score is obtained by reversing the scores on items 4, 5, 7, and 8, and then summing across all 10 items. Higher scores indicate higher perceived stress.
Change from baseline in depressive symptoms, as measured by the Patient Health Questionnaire - 9 scale, at 3 months post-intervention | Baseline and 3 months post-intervention
  The Patient Health Questionnaire - 9 (PHQ-9) is a 9-item scale used to assess the severity of depressive symptoms over the past two weeks and is based on Diagnostic and Statistical Manual (DSM- V) diagnostic criteria for major depression. Total scores range from 0 to 27, and clinical cut-points correspond to mild, moderate, moderately severe, and severe depression.
Change from baseline in pain catastrophizing, as measured by the Pain Catastrophizing Scale, at 3 months post-intervention. | Baseline and 3 months post-intervention
  The Pain Catastrophizing Scale (PCS) is a 13-item instrument which will evaluate the degree to which patients have negative self-statements and catastrophizing thoughts and ideations when in pain. The PCS uses a 5-point likert scale (0=not at all, 4=all the time) and consists of three subscales (rumination, magnification, helplessness).
Change from baseline in mindfulness, as measured by the Five Facet Mindfulness Questionnaire, at 3 months post-intervention. | Baseline and 3 months post-intervention
  Mindfulness will be measured using the Five Facet Mindfulness Questionnaire (FFMQ). The FFMQ is a 39-item instrument measuring five aspects of mindfulness: Non-reactivity to inner experience, observing, describing, acting with awareness, and non-judging of experience. Participants are asked to use a 5-point Likert-type scale (1 = never or rarely true 5 = very often or always true) to rate how true of them they believe each statement to be.
Change from baseline in quality of life, as measured by the Short-Form-12 Health Survey, at 3 months post-intervention. | Baseline and 3 months post-intervention
  Quality of life will be measured by the Short-Form-12 Health Survey (SF-12v.2). The SF-12v2 is a brief, twelve-item self-report measure based on the Short-Form-36. It includes items assessing eight health domains, such as bodily pain, social functioning, role limitations due to physical health, and general health perceptions. Two summary scores, the physical composite scale (PCS) and mental composite scale (MCS) are computed based on the 12 items. Scores range from 0 to 100, with higher scores indicating greater quality of life.
Change from baseline in quality of life, as measured by the Neuropathy-Specific Quality of Life Questionnaire (NeuroQOL). | Baseline and 3 months post-intervention
  The NeuroQoL was designed for and validated in patients with diabetic peripheral neuropathy and it captures the key dimensions of the patient's experience. Factor analysis revealed 3 physical symptom measures and 2 psychosocial functioning measures with good reliability (α = 0.86 - 0.95). This instrument was more strongly associated with severity of DPN than the SF-12 and more fully mediated the relationship between DPN and overall quality of life.
Change from baseline in quality of health and life, as measured by the The Summary of Diabetes Self-Care Activities (SDSCA). | Baseline and 3 months post-intervention
  The SDSCA is an 11-item self-report measure used to assess the diet, exercise, smoking, blood glucose testing and footcare habits of patients with diabetes. The scale has been found to be valid with moderate test-retest reliability.
Change from baseline in adverse reactions as a result of their glycemic control, as measured by the Blood Sugar Reactions Questionnaire. | Baseline and 3 months post-intervention
  These 5 questions were developed using the "Diabetes Care Profile" from the Michigan Diabetes Research and Training Centre as a guide.
Change from pre-intervention in biomarkers of stress, as measured by hair cortisol levels, at 3 months post-intervention. | Baseline and 3 months post-intervention
  Cortisol is a useful biomarker of stress levels. One cm hair samples will allow us to collect data on cortisol exposure over the past month. Hair cortisol will allow us to explore the relationship between systemic exposure to a potential mediator of the interaction between pain, stress, and glucose control in patients with diabetes. This novel aspect of the present proposal may help validate an important biomarker for investigating the neuro-endocrine correlates of chronic pain.
Change from baseline in glycemic control, as measured by blood levels of Hemoglobin A1c. | Baseline and 3 months post-intervention
  Blood samples will be obtained from participants and the measurement of Hemoglobin A1c performed. The concentrations Hemoglobin A1c will be quantified and recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Howard Nathan, MD, Principal Investigator — Ottawa Hospital Research Institute
Locations (1):
- The Ottawa Hospital, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Nathan HJ, Poulin P, Wozny D, Taljaard M, Smyth C, Gilron I, Sorisky A, Lochnan H, Shergill Y. Randomized Trial of the Effect of Mindfulness-Based Stress Reduction on Pain-Related Disability, Pain Intensity, Health-Related Quality of Life, and A1C in Patients With Painful Diabetic Peripheral Neuropathy. Clin Diabetes. 2017 Dec;35(5):294-304. doi: 10.2337/cd17-0077. PMID 29263572